CLINICAL TRIAL: NCT03435133
Title: Comparison of Prasugrel vs. Ticagrelor on Myocardial Injury in Revascularized ST Elevation Acute Myocardial Infarction Patients
Brief Title: Prasugrel vs. Ticagrelor on Myocardial Injury in STEMI
Acronym: COMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AORTICA Group (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, Head of Cardiology, PhD, MD, AORTICA Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARDIO2015.1
Record Dates: First submitted 2018-02-05; First posted 2018-02-15 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Primary angioplasty; Prasugrel; Ticagrelor; STEMI; cardiac magnetic resonance; infarct size; infarct injury
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prasugrel (Active Comparator)
  Interventions: Drug: Prasugrel
- Ticagrelor (Active Comparator)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — 60 mg oral bolus plus oral 10 mg once daily
  Arms: Prasugrel
Drug: Ticagrelor — 180 mg oral bolus plus oral 90 mg every 12 hours daily
  Arms: Ticagrelor

SUMMARY:
The investigators propose to perform a randomized clinical trial comparing prasugrel vs. ticagrelor in 60 patients with ST elevation acute myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention. The principal objective of the study would be analyzing the difference in myocardial infarction size measured by cardiac magnetic resonance at 6 months

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and one of the P2Y12 receptor inhibitors is the mainstay of treatment for patients with ST elevation acute myocardial infarction undergoing primary percutaneous coronary intervention. Prasugrel or ticagrelor have actually shown to be superior to clopidogrel improving the prognosis of these patients. However, the industrial interest has avoided any direct comparison between these two antiplatelets. Comparison is of great interest considering that only ticagrelor has shown to significantly reduce mortality. As ticagrelor may exert off-target effects through adenosine-related mechanisms, the investigators aimed to investigate whether ticagrelor reduces myocardial injury to a greater extent than prasugrel in patients with revascularized STEMI.

Patients with acute STEMI undergoing primary percutaneous coronary revascularization within 6 hours of chest pain, will be randomized to (1) prasugrel (a 60 mg oral loading and a 10-mg dailiy maintenance dose) or to (2) ticagrelor (a 180 mg loading dose and a 90 mg twice daily maintenance dose). The predefined primary end point is infarct sieze on magnetic resonance imaging at the end of the study (6 months). Magnetic resonance will be performed at day 1, day 7 and moth 6. Platelet reactivity, biomarkers and clinical outcomes will also be assesed.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older and equal or less than 75 years
* symptom onset within 12 hours before random assignment
* chest pain lasting more than 30 minutes
* ST-segment elevation of at least 0.1 mV in at least 2 limb leads, ST-segment elevation of at least 0.2 mV in 2 or more contiguous precordial leads, or left bundle-branch block or paced rhythm
* time from symptoms onset to randomization less than 6 hours
* no severe heart failure (Killip class <3)
* informed, written consent

Exclusion Criteria:

* history of myocardial infarction with Q wave
* history of surgical or percutaneous coronary revascularization
* cardiogenic shock, defined as a systolic blood pressure <90 mm Hg with no response to fluid administration or <100 mm Hg in patients with supportive treatment and no bradycardia
* history of stroke
* history of bronchial asthma
* symtomatic sinusal bradicardia or advance AV block
* history of hypersensitivity to aspirin, prasugrel or ticagrelor or contraindication to the doses established in the study
* patients pretreated with 600 mg of clopidogrel or more
* contraindication for the use of gadolinium during the magenitc resonance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Infarct size | 6 months
  Cardiac magnetic resonance imaging-assessed infarct size of left ventricular mass (%)

SECONDARY OUTCOMES:
Infarct size | up to two weeks
  Cardiac magnetic resonance imaging-assessed infarct size of left ventricular mass (%)
Myocardial salvage index | up to two weeks
  Cardiac magnetic resonance imaging-assessed myocardial salvage index
Microvascular obstruction | up to two weeks
  Cardiac magnetic resonance imaging-assessed microvascular obstruction
MACE | 6 months
  The rate of MACE defined as the composite of death, reinfarction, new-onset heart failure, or rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Sanchez, MD, PhD, Principal Investigator — Hospital Universitario Salamanca
Locations (1):
- Pedro Dorado, Salamanca, Spain